



## **INFORMED CONSENT FORM - Version 1.4 27/11/23**

Research Study Title: A cross-sectional study assessing the agreement between sonographer based assessment of the fatty liver using conventional ultrasound and attenuation imaging scoring.

| attenuation imaging | | | | |
|---|---|---|---|---|
| Participant Identification Number: | | Site: Bronglais Hospital, Aberystwyth | | ystwyth |
| Resea<br>Resea | Three copies will be made for: (1) Parcher, (3) Medical records (if relevant). rch Team Lead: Laura Mundy | | | · |
| | carefully the following statements a | Number:<br>and, if you agree, | 01970<br>please INITIAL (do | 635682<br>not tick) the |
| adjace | ent boxes. | | | INITIAL BOX |
| 1. | I confirm that I have read and unders – (Version 1.4 27/11/23) for the abopportunity to ask questions, and I are | oove research stud | y. I have had the | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected. | | | |
| 3. | If relevant, I understand that sections of any of my medical notes may be looked at by: responsible individuals from the Research Team or regulatory authorities where it is relevant to my taking part in research and the sponsor's representatives in Hywel Dda University Health Board for monitoring the conduct of the study. I give permission for these individuals to have access to my records. | | | |
| 4. | I confirm that I have understood all the above mentioned aspects and I agree to take part in the US & Attenuation imaging research study. | | | |
| or post | wish to receive a copy of the research<br>ed to you if you would prefer. Please of<br>be sent to. | | | |
| Email | | | | |
| Posta | al Address: | | | |
| Full Name of Participant (PRINT) | | Date: | Signature: | |
| Full N<br>(PRIN | Name of Person receiving consent<br>NT) | Date: | Signature: | |